CLINICAL TRIAL: NCT01179555
Title: Confronting Unequal Eye Care in Pennsylvania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Thomas Jefferson University (Other); Temple University (Other)
Responsible Party: Principal Investigator, Julia Haller, Ophthalmologist-in-Chief, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CURE-1837
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Diabetic Retinopathy; Diabetes Mellitus, Type 2; Glaucoma
Keywords: Diabetic Complications; Intervention Studies; African Americans; Vision Screening; Vision, Low; Geriatric Assessment; Outcomes Assessment; Cultural Characteristics; Cultural Competency; Appointment Adherence; Cost-effectiveness; Personalization of care; Follow-up Care
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus, Type 2; Glaucoma; Diabetes Complications; Vision, Low | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pt. 1 Behavioral Activation (Experimental): Behavioral Activation (BA) is a behavioral technique to help people overcome avoidant tendencies through goal setting, activity scheduling, and graded task assignment. The key component of BA involves developing an "Action Plan", and having the subject document each step of the plan as he or she implements it, reinforcing the steps towards goal attainment. "Action Plans" are easily applied to diabetes self-care tasks because the latter lend themselves to documentation of simple, step-by-step plans. In this study, a Community Health Educator (CHE) - interventionist will schedule and deliver four 45-60 minute in-home BA sessions within 3 months of randomization (i.e., one session every 2-3 weeks).
  Interventions: Behavioral: Behavioral Activation
- Pt. 1 Supportive Therapy (Placebo Comparator): The purpose of Supportive Therapy (ST) is to explore the impact of aging and diabetes on the subject's life. In contrast to the BA intervention, the interventionist does not discuss the importance of dilated eye exams. In subsequent sessions, ST facilitates and deepens knowledge about the subject's life situation in relation to his or her health and other life difficulties. The ST therapist encourages this process and creates an accepting, nondirective, and supportive opportunity for discussion.
  Interventions: Behavioral: Supportive Therapy

INTERVENTIONS:
Behavioral: Behavioral Activation — Baseline assessment plus 4 in-home problem solving therapy sessions.
  Other Names: BA - abbreviation
  Arms: Pt. 1 Behavioral Activation
Behavioral: Supportive Therapy — Baseline assessment plus 4 in-home sessions of supportive therapy.
  Other Names: ST-abbreviation
  Arms: Pt. 1 Supportive Therapy

SUMMARY:
Pt. 1 Diabetic retinopathy is a common eye condition among diabetic adults and can lead to severe vision impairment and even blindness. African Americans are more likely to have vision loss from diabetic retinopathy due to a variety of factors, including cultural barriers to care. The investigators aim to increase the rates of eye exams in diabetic African American adults by providing culturally relevant home-based interventions. These interventions will increase the knowledge about diabetes and the eyes and the awareness of ocular risks due to diabetes.

206 African American adults, over the age of 65, with diabetes will be recruited from primary care clinics at Thomas Jefferson and Temple University. Eligible patients who consent to participate will have baseline information taken about medical and ocular history, understanding of diabetes and a hemoglobin A1C level obtained. The subjects will then be randomized to one of two treatment conditions: Behavioral Activation or Supportive Therapy, each of which will be delivered over 4 sessions. Behavioral Activation will consist of educational materials, referral assistance for eye clinics, and addressing patient specific barriers to care. Supportive Therapy will consist of supportive but non-directional interaction with the patient exploring the impact of aging and diabetes on the patient's life. The investigators hypothesize that more patients who receive Behavioral Activation will have a dilated fundus exam (the primary outcome variable), understand the risks of diabetic complications and feel less depression then subjects who receive Supportive Therapy.

DETAILED DESCRIPTION:
An additional aim was added to this project, examining the effect of a telephone intervention on eye care adherence and comparing the efficacy of the intervention to usual care and automated telephone screenings.

Glaucoma is a group of chronic, neurodegenerative diseases of the optic nerve, which leads to an increase in intraocular pressure, gradual changes in the visual field (VF), and progressive vision loss. Glaucomatous vision loss is preventable with proper eye care, including adherence to follow-up appointments and medications. Interventions that improve appointment adherence have the potential to prevent more severe glaucomatous disease. The primary purpose of this study is to determine the efficacy of a multifaceted intervention system, which includes a customized letter and personal telephone outreach, in improving appointment adherence in patients with glaucoma. In order to improve strategies to reduce the rate of appointment non-adherence, shared characteristics of adherent versus non-adherent patients with glaucoma will be identified and compared to patient characteristics in the previous literature. A secondary goal of this study is to analyze the cost-effectiveness of this multifaceted intervention on appointment adherence in patients with glaucoma.

ELIGIBILITY:
Pt. 1

Inclusion Criteria:

* African-American race (self-identified)
* Age ≥ 65 years
* Type II Diabetes Mellitus (physician diagnosis) for at least 1 year
* No medical documentation of a DFE by an ophthalmologist or an optometrist within the past 12 months
* Self-report of no DFE within the past 12 months

Exclusion Criteria:

* Cognitive Impairment (Mini-Mental Status Examination ≤ 24)
* Current clinically significant psychiatric disorder other than depression
* Current medical disorder that limits life expectancy (≤ 12 months) or need for dialysis
* Hearing impairment that precludes research participation

Pt. 2

Inclusion Criteria:

* Glaucoma (physician diagnosis)
* Scheduled for a follow-up appointment that meets the American Academy of Ophthalmology (AAO) follow-up guidelines
* Attended the Wills Eye Glaucoma Clinic from September 1, 2012 to October 31, 2013
* Age ≥ 21 years old
* Able to understand and speak English

Exclusion Criteria:

* Diagnosed with a pre-existing medical condition that would preclude the subject from providing reliable and valid data
* Individual was asked to follow-up in less than a month.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2010-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pt. 1 Dilated Fundus Exam (DFE) | 6-month follow-up assessment
  At the 6-month follow-up assessment, patients will be asked if they got a dilated fundus exam since the baseline assessment. If a DFE is self-reported, it will be confirmed by ophthalmology chart review

SECONDARY OUTCOMES:
Pt. 1 Risk perceptions of diabetes | 6-month follow up assessment
  Risk Perception Survey-Diabetes Mellitus (RPS-DM) has 5 subscales:
  1) Personal Control, 2) Optimistic Bias, 3) Personal Disease Risk, 4) Comparative Environmental Risk, 5) Risk Knowledge
Pt. 1 Diabetes self-care behaviors | 6-month follow up assessment
  Yields a global scale that summarizes self-care behaviors
Pt. 1 Depressive Symptoms | 6-month follow up assessment
  Patient Health Questionnaire-9 (PHQ-9)
Pt. 2 Appointment Adherence Characteristics | Dependent on Diagnosis
  To assess the relationship between appointment adherence and particular demographic characteristics, clinical factors, and systems-level variables.

OTHER OUTCOMES:
Pt. 2 Cost-effectiveness | Conclusion of Study
  To determine which aspects of the intervention are most costly, and whether these aspects can be delivered more efficiently in order to promote broader translation.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Haller, MD, Principal Investigator — Wills Eye; Lisa Hark, PhD, RD, Study Director — Wills Eye
Locations (3):
- United States (3):
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Wills Eye Health System, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Several manuscripts have been published.

REFERENCES:
- [Background] Weiss DM, Casten RJ, Leiby BE, Hark LA, Murchison AP, Johnson D, Stratford S, Henderer J, Rovner BW, Haller JA. Effect of Behavioral Intervention on Dilated Fundus Examination Rates in Older African American Individuals With Diabetes Mellitus: A Randomized Clinical Trial. JAMA Ophthalmol. 2015 Sep;133(9):1005-12. doi: 10.1001/jamaophthalmol.2015.1760. PMID 26068230
- [Background] Rovner BW, Haller JA, Casten RJ, Murchison AP, Hark LA. Cultural and Cognitive Determinants of Personal Control in Older African Americans with Diabetes. J Natl Med Assoc. 2015 Jun;107(2):25-31. doi: 10.1016/S0027-9684(15)30021-3. Epub 2015 Dec 2. PMID 27269487
- [Derived] Pizzi LT, Tran J, Shafa A, Waisbourd M, Hark L, Murchison AP, Dai Y, Mayro EL, Haller JA. Effectiveness and Cost of a Personalized Reminder Intervention to Improve Adherence to Glaucoma Care. Appl Health Econ Health Policy. 2016 Apr;14(2):229-40. doi: 10.1007/s40258-016-0231-8. PMID 26924099